CLINICAL TRIAL: NCT05982730
Title: SegwayPD: The Effect of Sensory-augmented Postural Training Using Segway on Motor and Cognitive Function in Individuals With Parkinson's Disease
Acronym: SegwayPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Yasin Dhaher, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 46179; STU-2023-0066
Record Dates: First submitted 2023-07-06; First posted 2023-08-09 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD - individuals with Parkinson Disease, either male or female (Experimental): Individuals, aged 50-85, with a clinical diagnosis of idiopathic Parkinson Disease, either male or female, with moderate disease stage presenting balance alterations (Hoehn or Yahr stage III)
  Interventions: Behavioral: Sensory-Augmented Postural Training

INTERVENTIONS:
Behavioral: Sensory-Augmented Postural Training — To examine the safety and efficacy of postural training emphasized on the integration of multiple sensory information into motor control and to assess the effectiveness of postural training using Segway

SUMMARY:
The purpose of this study is to examine the safety and efficacy of postural training emphasized on the integration of multiple sensory information into motor control in individuals with PD. This project is a proof-of-concept study to assess the effectiveness of postural training using Segway, which serves a platform to provide augmented and continuous proprioceptive and visuospatial information during postural training.

DETAILED DESCRIPTION:
The purpose of this study is to examine the safety and efficacy of postural training emphasized on the integration of multiple sensory information into motor control in individuals with PD (Parkinson's disease). This project is a proof-of-concept study to assess the effectiveness of postural training using Segway, which serves a platform to provide augmented and continuous proprioceptive and visuospatial information during postural training. Specifically, we will measure postural sway during quiet standing, single and dual-task walking performances, and brain activation during single and dual-task walking from the regions involved in planning and execution of locomotion; these include dorsolateral prefrontal cortex, premotor cortex and primary motor cortex. The changes in visuospatial function and proprioception after training will also be assessed. Individuals with moderate disease stage of PD exhibiting postural instability will be recruited. The participants will receive 1-week training and be assessed at 3 time points: 1-week before, before, and after the training.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of idiopathic PD with moderate disease stage presenting balance alterations (Hoehn and Yahr stage III)
* being stable on medication for at least 1 month
* the ability to stand and walk unsupported for 5 min both on and off medication
* age between 50 and 85

Exclusion Criteria:

* neurological disorders other than PD
* major unstable medical illnesses
* sensory or musculoskeletal disorders (e.g., diabetes, uncorrected visual problems, arthritis, severe hearing impairments) that will prohibit the ability to perform the assessment tests and receive training

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline postural sway at week 3 | Week 1 (2 assessments), Week 3 (1assessment)
  The midpoint between the tip of left and right calcaneus bones is considered as the origin of the reference system of the center of pressure (CoP). The CoP displacement along lateral and anterior-posterior axes are measured. The overall size of postural sways will be estimated from the ellipse area conveying 85% of the total CoP samples. The postural sway obtained from 2 assessments during week 1 will be averaged and used as baseline value. The postural sway obtained at week 3 is used to analyze the change from baseline due to training intervention (week 2).

SECONDARY OUTCOMES:
Feasibility of Segway training | Week 3 (1 assessment)
  The attendance of training session for each participant will be used to assess the feasibility of the 1-week postural training. Adherence above 80% will indicate that the participants receive the training well.
Change from baseline gait spatiotemporal parameters at week 3 | Week 1 (2 assessments), Week 3 (1assessment)
  Spatiotemporal parameters will be used to characterized walking in dual task and single task conditions. One gait cycle will be defined as period from heel strike to the consecutive heel strike of the ipsilateral leg. The gait's spatiotemporal parameters obtained from 2 assessments during week 1 will be averaged and used as baseline value. The gait's spatiotemporal parameters obtained at week 3 is used to analyze the change from baseline due to training intervention (week 2).
Change from baseline EEG spectral ratio at week 3 | Week 1 (2 assessments), Week 3 (1assessment)
  The absolute powers in delta (0.5-4 Hz), theta (4-8 Hz), alpha (8-13 Hz), and beta (13 - 30 Hz) frequency bands obtained using Fast Fourier Transform will be used to calculate the spectral ratio of the frequency bands. The spectral ratio is defined as ratio of the sum of absolute powers in the alpha and beta bands divided by the sum of the absolute power in the delta and theta frequency bands. The spectral ratio obtained from 2 assessments during week 1 will be averaged and used as baseline value. The spectral ratio obtained at week 3 is used to analyze the change from baseline due to training intervention (week 2).

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Dhaher, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States